CLINICAL TRIAL: NCT04545034
Title: After Effects of a Water Aerobics Session on Blood Pressure of Hypertensive Elderly: a Randomized Clinical Trial
Brief Title: Water Aerobics Session on Blood Pressure of Hypertensive Elderly.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Centro Universitário de Anapolis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PPGMHR-001/20
Record Dates: First submitted 2020-08-25; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Hypertension; Blood Pressure
Keywords: hypertension; water aerobic exercise; elderly; blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: This is a randomized crossover clinical trial carried out with 25 hypertensive women. The study procedures took place over three days with an interval of 48 hours, and included evaluation session, an experimental protocol (EP) and a control protocol (CP).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water aerobic exercise protocol (Experimental): Walter aerobic exercise session would be used to treat blood pressure in elderly hypertensive people.
  Interventions: Other: water aerobic exercise
- Control Group (No Intervention): No exercise intervention would be used.

INTERVENTIONS:
Other: water aerobic exercise — The EP would be formed by continuous session of dynamic water aerobic exercise which consisted of a dynamic warm-up period (5 minutes), an active exercise period at the established intensity of HR (35 minutes), and a cooldown period (5 minutes) to total 45 minutes, with a intensity of 75%HR.
  Arms: Water aerobic exercise protocol

SUMMARY:
This randomized controlled trial aimed to determine the subacute blood pressure effects of pharmacologically-treated elderly hypertensive patients after a single session of water aerobic exercise.

DETAILED DESCRIPTION:
A randomized clinical trial with a crossover design was conducted at an aquatic center and an exercise physiology laboratory. All subjects read and signed an informed consent form before participating in the study. Additionally, this study follows the recommendations as proposed by the CONSORT Statement.

The minimum sample size was determined based on a previous study conducted by our research group. We estimated a sample size of 24 individuals for a 5% significance level, power of 95%, and a 10 mmHg difference in systolic blood pressure (SBP). The inclusion criteria were age between 65 and 85 years; practice exercise (almost 3 days-week); use of anti-hypertensive drugs; systolic blood pressure (SBP) ≤160 mmHg and diastolic blood pressure (DBP) ≤100 mmHg documented by a physician. The exclusion criteria were body mass index (BMI) >35 kg/m2; decompensated diabetes mellitus and/or cardiac failure; active smoker; any febrile condition and/or infectious diseases; cardiovascular event in the 3 months preceding the study; hepatopathy; physical or mental limitations that prevent exercising.Participants were recruited using local media advertisement. The potential participants were asked to attend an on-site visit before the experiment. In this visit, the study procedures were explained and they those who agreed to participate signed an informed consent form. Then, they were interviewed using a questionnaire and information on medical history and symptoms among others was collected, and in sequence they underwent physical and medical evaluations with measurements (weight, height, BMI, BP).The included participants were then assigned to either the experimental protocol (EP) or the control protocol (CP) with 48 hours between sessions. Randomization was performed by digital system (www.randomization.org) at a 1:1 allocation ratio and participants were assigned to either exercise or control session. All sessions occurred at the same time (10 to 11 am) with 2 days between sessions.

The EP consisted of one water aerobic exercise session carried out at the aquatic center in a 1.4 m-deep swimming pool with water at an average temperature of 28.5°C, with a average air temperature of 30°C. The EP was a continuous session of dynamic water aerobic exercise which consisted of a dynamic warm-up period (5 minutes), an active exercise period at the established intensity of HR (35 minutes), and a cooldown period (5 minutes) to total 45 minutes. Heart rate (HR) was continuously measured with heart monitors (Polar, RS 800 CX®, USA) to confirm the intensity of the exercise. The EP intensity was calculated according to the formula proposed by Kruel et al. (2014) [27] for exercise in an aquatic. Besides, we used the Borg Rating of Perceived Exertion Scale to measure exercise intensity level in those participants on β-blockers, exercising around number 13 of the scale during active exercise. Water aerobic exercises included flexion, extension, abduction, and adduction of upper and lower limbs. It was a continuous session with no rest between.The CP was a 45-min session of no exercise. It was also held at the aquatic center in environment conditions similar to those of the exercise session. During this session, the participants remained seated or standing as desired, and were allowed to read, talk and drink water, but did nothing else.

Blood pressure was measured with the patient seated using an internationally validated semi-automatic BP monitor (Omron 705-CP, Matsusaka, Japan) following techniques adopted by The Seventh Report [1]. BP was measured before the session (Pre); immediately after (Min-0) and every 10 minutes until 60 minutes after the protocols had been performed (Min-10, Min-20, Min-30, Min-40, Min-50 and Min-60). The measurements were repeated at 2-minute intervals and the calculation of the mean of the two measurements.

ELIGIBILITY:
Inclusion Criteria:

* age between 65 and 85 years;
* practice exercise (almost 3 days-week);
* use of anti-hypertensive drugs;
* systolic blood pressure (SBP) ≤160 mmHg and diastolic blood pressure (DBP) ≤100 mmHg documented by a physician

Exclusion Criteria:

* body mass index (BMI) >35 kg/m2;
* decompensated diabetes mellitus and/or cardiac failure;
* active smoker;
* any febrile condition and/or infectious diseases;
* cardiovascular event in the 3 months preceding the study;
* hepatopathy;
* physical or mental limitations that prevent exercising.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 25 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Blood pressure after water aerobic exercise in elderly hipertensive | Baseline response to 10 days
  Blood pressure was measured with the patient seated using an internationally validated semi-automatic BP monitor (Omron 705-CP, Matsusaka, Japan) following techniques adopted by The Seventh Report [1]. BP was measured before the session (Pre); immediately after (Min-0) and every 10 minutes until 60 minutes after the protocols had been performed (Min-10, Min-20, Min-30, Min-40, Min-50 and Min-60). The measurements were repeated at 2-minute intervals and the calculation of the mean of the two measurements.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Centro Universitário de Anápolis - UniEVANGÉLICA, Anápolis, Goiás
  - Raphael Martins Da Cunha, Goiânia, Goiás

IPD SHARING:
Plan to Share IPD: No